CLINICAL TRIAL: NCT04753554
Title: Can Hyperoxia be Prevented With Noninvasive Monitoring in On-pump Cardiac Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ipek Bostancı, Specialist, MD, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2020-281
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Hyperoxia; Oxygen Reserve Index; Cardiac Surgery
Keywords: hyperoxia; ORI
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional group (Active Comparator): The patient group that whose oxygenation will be managed by blood gas analysis.
  Interventions: Device: ORI group; Other: Conventional group
- ORI group (Experimental): The patient group that whose oxygenation will be managed by ORI values
  Interventions: Device: ORI group

INTERVENTIONS:
Device: ORI group — The patient group whose oxygenation will be managed by ORI values. Hyperoxia or hypoxia will be prevented by using also blood gas analysis in critically ill patients.
Other: Conventional group — In this patient group oxygenation will be managed as usual, using blood gas analysis.
  Arms: Conventional group

SUMMARY:
In our study, we aimed to observe the usability of non-invasive monitoring methods in oxygenation management, using non-invasive monitoring techniques, preventing hyperoxia and avoiding oxidative damage-related complications in patients undergoing on-pump cardiac surgery.

DETAILED DESCRIPTION:
In on-pump cardiac surgery; The risk of organ perfusion disorders is high due to the heart-lung pump process they involve. It is essential to avoid hypoxia in such patient groups in order to prevent perfusion disorders. While preventing hypoxia, hyperoxia processes can be observed frequently in patients. In order to avoid complications related to hyperoxia and oxidative damage, oxygenation management should be followed closely. Today, non-invasive monitoring methods are being used in this field. In our study, we aimed to observe the usability of this method in oxygenation management and avoidance of hyperoxia by performing oxygenation management over ORI (oxygene reserve index) value using the Masimo Root + Radical 7 Rainbow SET device with SPHB finger probe.

30 patients will bi included in our study; and they will be divided into two groups: In one group oxygenation management will be performed by conventional method, such as blood gas analysis. In other group ORI values will be used to manage oxygenation. Lung ultrasound will be performed in both groups to see if there will be any sign for atelectasis, preoperatively and postoperatively.

Kidney and liver functions will also be investigated before and after surgery. For cognitive disfunction evaluation; CAM-ICU scores will be recorded in both groups at 24 hours after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 - 75
* Patients undergoing on-pump cardiac surgery

Exclusion Criteria:

* Patients with advanced CHF (EF <40%)
* Patients with advanced COPD (FEV1 <60%)
* Patients with a history of CVD
* Patients with advanced carotid lesions (> 50-70% of stenosis)
* Patients with renal failure
* Patients with liver failure
* Patients with cardiac arrhythmia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 24 hours
  This will be measured preoperatively; routinely 4 times perioperatively, if there is any intervention after the intervention; and 3 times postoperatively. Reported as % (T1: Preoperative, T2: after intubation, T3: aortic cross clemp o, T4: aortic cross clemp off, T5: After decanullation; T6: 2 hours after operation; T7: After extubation; T8: 24 hours after operation)
Parsial oxygen pressure | 24 hours
  This will be measured preoperatively by blood gas analysis; routinely 4 times perioperatively, if there is any intervention after the intervention; and 3 times postoperatively. Reported as mmHg. (T1: Preoperative, T2: after intubation, T3: aortic cross clemp o, T4: aortic cross clemp off, T5: After decanullation; T6: 2 hours after operation; T7: After extubation; T8: 24 hours after operation)
Oxygen reserve index | 6 hours
  This will be measured only in ORI group patients using Masimo device preoperatively; routinely 4 times perioperatively and if there is any intervention after the intervention. (T1: Preoperative, T2: after intubation, T3: aortic cross clemp o, T4: aortic cross clemp off, T5: After decanullation)

SECONDARY OUTCOMES:
Lactate levels | 24 hours
  This will be measured by blood gas analysis; preoperatively; routinely 4 times perioperatively, if there is any intervention after the intervention; and 3 times postoperatively. (T1: Preoperative, T2: after intubation, T3: aortic cross clemp o, T4: aortic cross clemp off, T5: After decanullation; T6: 2 hours after operation; T7: After extubation; T8: 24 hours after operation)
Near-infrared Spectroscopy values (Left/Right) | 24 hours
  This will be measured using Masimo device; preoperatively; routinely 4 times perioperatively, if there is any intervention after the intervention; and 1 time postoperatively. T1: Preoperative, T2: after intubation, T3: aortic cross clemp o, T4: aortic cross clemp off, T5: After decanullation; T8: 24 hours after operation)
Urine & Creatinine & ALT & AST | 24 hours
  This will be measured using blood analysis preoperatively and postoperatively. (T1: Preoperative; T8: 24 hours after operation)
Lung Ultrasound Scores | 24 hours
  This will be measured by using ultrasound device preoperatively and postoperatively. (T1: Preoperative; T8: Postoperative)
CAM-ICU | 24 hours
  This will be measured by examination of patient postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy / Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No